CLINICAL TRIAL: NCT06648135
Title: a Novel Socket Evaluation System and Its Impact on Bone Formed Labial to Bone Immediate Anterior Implants. A 1-year Clinical Trial.
Brief Title: Labial Bone Thickness Around Immediate Implants in the Esthetic Zone Following a Novel Socket Evaluation System
Status: Not yet recruiting | Type: Observational
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Exectutive and Clinical director of Implantology Master program, MIU, Misr International University
Other Study IDs: IDCE 14
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Immediate Implant Placement
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone grafts: Immediate implant placed with bone grafts in the labial gap
  Interventions: Procedure: Immediate implants with bone grafts
- No bone grafts: Immediate implant placed without bone grafts or any grafting substitutes in the labial gap
  Interventions: Procedure: Immediate implant placed without bone grafts or any grafting substitutes in the labial gap

INTERVENTIONS:
Procedure: Immediate implants with bone grafts — Immediate implants with bone grafts
  Groups: Bone grafts
Procedure: Immediate implant placed without bone grafts or any grafting substitutes in the labial gap — Immediate implant placed without bone grafts or any grafting substitutes in the labial gap
  Groups: No bone grafts

SUMMARY:
The anterior maxilla is a particularly challenging area for immediate implant placement due to its thin buccal bone walls. These walls are more susceptible to resorption after tooth extraction, which can lead to significant bone loss and inadequate support for an implant. However, Different socket dimension may affect the amount of bone formed labial to the implant, regardless of the garfting procedure.

DETAILED DESCRIPTION:
Bone formation labial to the immediate implant is not related to the initial thick- ness of the labial plate of bone, rather than the initial labio-palatal socket dimension. this study aims to evaluate the bone formed labial to the implant following a Novel Socket Evaluation System.

ELIGIBILITY:
Inclusion Criteria:

* Immedaite implants in anterior maxilla
* thick gingival phenotype
* intact but thin labial plate of bone (≤1mm)
* sufficient apical bone to attain implant primary stability (a minimum of 35 Ncm insertion torque)

Exclusion Criteria:

* smokers
* pregnant women
* patients with systemic disease
* patients with parafunctional habits such as bruxism or clenching,
* infected socket
* periapical pathosis
* history of radiotherapy or chemotherapy within the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Bone labial to the implant | one year
  measured at three levels 0, 2, and 5 mm below the labial bone crest after one year. Using fusion software.

SECONDARY OUTCOMES:
Bone area at the Interproximal component | preoperative
  Bone area at the mesial and distal Interproximal component in mm2

CONTACTS AND LOCATIONS:
Locations (1):
- International Dental Clinic Educational centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No